CLINICAL TRIAL: NCT02068235
Title: Single-center, Open-label, Randomized, Two-way Crossover Study to Investigate the Absolute Bioavailability of a Single Oral Dose of Ponesimod in Healthy Male Subjects
Brief Title: Study to Investigate the Absolute Bioavailability of a Single Oral Dose of Ponesimod in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AC-058-114
Record Dates: First submitted 2014-02-19; First posted 2014-02-21 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Healthy
Keywords: Ponesimod; Bioavailability; Pharmacokinetics; Safety
MeSH Terms: interventions — ponesimod; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pilot Phase (Experimental): Subjects will receive a single intravenous (i.v.) dose of 5 mg ponesimod dissolved in 50 mL sterile 0.9% sodium chloride (NaCl) solution as a 3-hour infusion in the fasted state in the morning (infusion rate: 0.028 mg/min).
  Interventions: Drug: Ponesimod 5mg i.v.
- Treatment A/Treatment B (Experimental): Subjects will receive Treatment A followed by Treatment B.
  Treatment A: a single i.v. dose of ponesimod administered in the fasted state in the morning.
  Treatment B: a single oral dose of ponesimod (10 mg) administered as 1 tablet in the fasted state in the morning.
  There will be a washout period between doses of 12-15 days.
  Interventions: Drug: Ponesimod i.v.; Drug: Ponesimod 10 mg tablet
- Treatment B/Treatment A (Experimental): Subjects will receive Treatment B followed by Treatment A.
  Treatment A: a single i.v. dose of ponesimod administered in the fasted state in the morning.
  Treatment B: a single oral dose of ponesimod (10 mg) administered as 1 tablet in the fasted state in the morning.
  There will be a washout period between doses of 12-15 days.
  Interventions: Drug: Ponesimod i.v.; Drug: Ponesimod 10 mg tablet

INTERVENTIONS:
Drug: Ponesimod 5mg i.v.
  Arms: Pilot Phase
Drug: Ponesimod i.v. — Dose and infusion rate will be adjusted according to the results of the pilot phase
  Arms: Treatment A/Treatment B; Treatment B/Treatment A
Drug: Ponesimod 10 mg tablet
  Arms: Treatment A/Treatment B; Treatment B/Treatment A

SUMMARY:
This study consists of a single-dose pilot phase and a randomized, two-way crossover, single-dose main phase.The aim of this study is to evaluate the absolute bioavailability of the oral formulation (tablet) of ponesimod compared to an intravenous (i.v.) ponesimod formulation. Three subjects will be included in the pilot phase and 12 subjects in the main crossover phase.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in the local language prior to any study-mandated procedure.
* Body mass index ≥ 18 and ≤ 28 kg/m^2 at screening.
* No clinically significant findings on the physical examination at screening.
* Systolic blood pressure (SBP) 100-145 mmHg and diastolic blood pressure (DBP) 50-90 mmHg, measured on the dominant arm, after 5 min in the supine position at screening and Day -1 of pilot phase/ first treatment period in main phase.
* 12-lead ECG without clinically relevant abnormalities at screening and Day -1 pilot phase / first treatment period in main phase.
* Negative results from urine drug screen at screening and Day -1 pilot phase / first treatment period in main phase.
* Hematology and clinical chemistry variables not deviating from the normal range to a clinically relevant extent at screening.
* Ability to communicate well with the investigator, in the local language, and to understand and comply with the requirements of the study.

Exclusion Criteria:

* Known allergic reactions or hypersensitivity to the active compound or any excipients of the drug formulation(s).
* History or clinical evidence of any disease and/or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism, or excretion of the study drug (appendectomy and herniotomy allowed, cholecystectomy not allowed).
* Veins unsuitable for i.v. puncture on either arm (e.g., veins that are difficult to locate, access, or puncture or veins with a tendency to rupture during or after puncture).
* Heart rate < 50 or > 95 beats per minute (bpm) at screening or Day -1 of pilot phase / first treatment period in main phase on 12-lead ECG measured after 5 min in the supine position.
* PR interval (time interval from the beginning of the P wave to the beginning of the QRS complex) > 200 ms at screening and Day -1 of pilot phase / first treatment period in main phase.
* Subjects with personal or family history of long QT (time interval from beginning of the Q wave until end of the T wave) syndrome or hypokalemia.
* Previous history of fainting, collapse, syncope, orthostatic hypotension, or vasovagal reactions.
* Previous exposure to the study medication within 3 months prior to screening.
* Any immunosuppressive treatment within 6 weeks or 5 half-lives of the drug, whichever is longer, before study drug administration.
* Treatment with another investigational drug within 3 months or 10 half-lives of the drug, whichever is longer, prior to screening or participation in more than 4 investigational drug studies within 1 year prior to screening.
* History or clinical evidence of alcoholism or drug abuse within the 3-year period prior to screening.
* Excessive caffeine consumption, defined as ≥ 800 mg (7 cups of coffee or 14 cups of tea) per day at screening.
* Smoking within the last 3 months prior to screening and inability to refrain from smoking during the course of the study.
* Treatment with any prescribed medications (including vaccines) or over-the-counter (OTC) medications (including herbal medicines) within 2 weeks prior to screening.
* Loss of 250 mL or more of blood within 3 months prior to screening.
* Lymphopenia (< 1000 cells/μL) at screening or Day -1 of pilot phase / first treatment period in main phase.
* Viral, fungal (with exception of onychomycosis and dermatomycosis), bacterial, or protozoal infection within 4 weeks before the first study drug administration.
* Positive results from the hepatitis serology, except for vaccinated subjects or subjects with past but resolved hepatitis, at screening.
* Positive results from the human immunodeficiency virus (HIV) serology at screening.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.
* Legal incapacity or limited legal capacity at screening.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC(0-144h)) of ponesimod | 7 Days
  Blood samples for pharmacokinetic analysis will be taken immediately prior to dosing with ponesimod, and at various time points up to 7 days after dosing. AUC(0-144) will be calculated according to the linear trapezoidal rule using the measured concentration-time values above the limit of quantification.
Area under the plasma concentration-time curve (AUC(0-infinity)) of ponesimod | 7 Days
  Blood samples for pharmacokinetic analysis will be taken immediately prior to dosing with ponesimod, and at various time points up to 7 days after dosing. AUC(0-infinity) will be calculated by combining AUC(0-144) and AUC(extra). AUC(extra) represents an extrapolated value obtained by Ct/λz, where Ct is the last plasma concentration measured above the limit of quantification and λz represents the terminal elimination rate constant determined by log-linear regression analysis of the measured plasma concentrations of the terminal elimination phase.
Maximum plasma concentration (Cmax) of ponesimod | 7 Days
  Blood samples for pharmacokinetic analysis will be taken immediately prior to dosing with ponesimod, and at various time points up to 7 days after dosing. Cmax will be calculated on the basis of the blood sampling time points.
Plasma half life (t1/2) of ponesimod | 7 Days
  Blood samples for pharmacokinetic analysis will be taken immediately prior to dosing with ponesimod, and at various time points up to 7 days after dosing. t1/2 will be calculated on the basis of the blood sampling time points.
Time to maximum plasma concentration (tmax) after oral administration of ponesimod | 7 Days
  Blood samples for pharmacokinetic analysis will be taken immediately prior to dosing with ponesimod, and at various time points up to 7 days after dosing. tmax will be calculated on the basis of the blood sampling time points.
Total body clearance (CL) after intravenous administration of ponesimod | 7 Days
  Blood samples for pharmacokinetic analysis will be taken immediately prior to dosing with ponesimod, and at various time points up to 7 days after dosing. CL Total body clearance will be calculated as follows: CL = Dose / AUC(0-infinity).
Volume of distribution (Vss) after intravenous administration of ponesimod | 7 Days
  Blood samples for pharmacokinetic analysis will be taken immediately prior to dosing with ponesimod, and at various time points up to 7 days after dosing. Vss will be estimated by CL [(AUMC/AUC) - (infusion time/2)], where AUMC is the area under the first moment curve.
Absolute bioavailability (F) of after oral administration of ponesimod | 7 Days
  Blood samples for pharmacokinetic analysis will be taken immediately prior to dosing with ponesimod, and at various time points up to 7 days after dosing. F will be calculated using the geometric means (as derived by the mixed effect model) of AUC(0-infinity).

SECONDARY OUTCOMES:
Change from baseline up to Day 7 in systolic blood pressure | 7 Days
  Blood pressure (systolic and diastolic) and pulse rate will be measured using an automatic oscillometric device, always on the leading arm (i.e., leading arm = writing arm). Measurements will be recorded in the supine position after the subject has rested for a 5-minute period.
Change from baseline up to Day 7 in diastolic blood pressure | 7 Days
  Blood pressure (systolic and diastolic) and pulse rate will be measured using an automatic oscillometric device, always on the leading arm (i.e., leading arm = writing arm). Measurements will be recorded in the supine position after the subject has rested for a 5-minute period.
Change from baseline up to Day 7 in pulse rate | 7 Days
  Blood pressure (systolic and diastolic) and pulse rate will be measured using an automatic oscillometric device, always on the leading arm (i.e., leading arm = writing arm). Measurements will be recorded in the supine position after the subject has rested for a 5-minute period.
Change from baseline up to Day 7 in heart rate | 7 Days
  Heart rate will be determined from standard 12-lead electrocardiographs (ECGs) recorded in the supine position, after a 5-minute period of resting.
Change from baseline up to Day 7 in PR interval (time interval from the beginning of the P wave to the beginning of the QRS complex) | 7 Days
  PR interval will be determined from standard 12-lead electrocardiographs (ECGs) recorded in the supine position, after a 5-minute period of resting.
Change from baseline up to Day 7 in QRS duration (time interval from the beginning of the Q wave to the end of the S wave) | 7 Days
  QRS duration will be determined from standard 12-lead electrocardiographs (ECGs) recorded in the supine position, after a 5-minute period of resting.
Change from baseline up to Day 7 in QT interval (time interval from beginning of the Q wave until end of the T wave) | 7 Days
  QT interval will be determined from standard 12-lead electrocardiographs (ECGs) recorded in the supine position, after a 5-minute period of resting.
Change from baseline up to Day 7 in QT interval according to Bazett's correction (QTcB) | 7 Days
  QTcB interval will be determined from standard 12-lead electrocardiographs (ECGs) recorded in the supine position, after a 5-minute period of resting. The QTcB interval is the QT interval (interval from beginning of the Q wave until end of the T wave) corrected for heart rate with Bazett's formula (QTcB = QT/RR^0.5 where RR is 60/heart rate)
Change from baseline up to Day 7 in QT interval according to Fridericia's correction (QTcF) | 7 Days
  QTcF interval will be determined from standard 12-lead electrocardiographs (ECGs) recorded in the supine position, after a 5-minute period of resting.The QTcF interval is the QT interval (interval from beginning of the Q wave until end of the T wave) corrected for heart rate with Fridericia's formula (QTcB = QT/RR^0.33 where RR is 60/heart rate)
Frequency of treatment-emergent ECG abnormalities from up to Day 7 | 7 Days
  Treatment-emergent abnormalities will be determined from standard 12-lead ECGs recorded in the supine position, after a 5-minute period of resting. Treatment-emergent ECG abnormalities are any ECG abnormalities that occur up to 144 hours after each study drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Baldoni, PharmD, PhD, Study Director — Actelion
Locations (1):
- Simbec Research Limited, Merthyr Tydfil, United Kingdom